CLINICAL TRIAL: NCT03869281
Title: Effect of Type 1 Diabetes Remission by Pancreas Transplantation Alone on Fracture Risk: a Retrospective Matched Cohort Study
Brief Title: Fracture Risk After Pancreas Transplantation (FraPaT)
Acronym: FRAPAT
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Caterina Conte, Assistant Professor, Università Vita-Salute San Raffaele
Other Study IDs: FRAPAT; 155/INT/2018 (Other: Ethics Committee)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1; Fractures, Bone
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Fractures, Bone | interventions — Pancreas Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTA: patients who underwent their first deceased donor PTA, or second deceased donor PTA if their first graft was explanted within a week, at the IRCCS San Raffaele Hospital between 2 January 2005 and 31 December 2017
  Interventions: Procedure: Pancreas transplantation alone
- Controls: outpatients with T1D attending the Endocrinology Unit at IRCCS San Raffaele Hospital and patients listed for a first deceased donor PTA

INTERVENTIONS:
Procedure: Pancreas transplantation alone — Pancreas transplantation
  Groups: PTA

SUMMARY:
Individuals with type 1 diabetes (T1D) are at greater risk of fracture than non-diabetic subjects. Although the mechanisms underlying bone fragility in T1D are not completely understood, insulin deficiency seems to play a key role.

To date, no information is available on the effect of diabetes remission after pancreatic transplantation alone (PTA) on the risk of fractures in T1D individuals with preserved kidney function.

The overall objective of this retrospective cohort study is to evaluate the effect of T1D remission after PTA on fracture risk.

The primary endpoint will be the difference in fracture incidence (any fracture) between the PTA group and the control group. For the PTA group, the incidence of fractures after transplantation will be considered.

Data from patients who underwent PTA at IRCCS San Raffaele Hospital from January 2, 2005 to December 31, 2017 will be compared with age-, gender- and disease duration-matched controls from the pool of outpatients with T1D attending the Endocrinology Unit at the same Institution. Anthropometric, anamnestic, laboratory data and data on the history of fractures and past/current therapies will be collected.

With this study, for the first time we will be able to obtain information on the effects of diabetes remission on the risk of fracture. We expect that the remission of diabetes will result in a beneficial effect on the fracture risk.

ELIGIBILITY:
Inclusion Criteria (PTA group)

* T1D patients who received their first PTA, or second PTA only if their first graft was explanted within a week, between 2 January 2005 and 31 December 2017
* age ≥18 and < 65 years
* willingness to participate in this observational study

Inclusion Criteria (control group)

* Type 1 diabetes
* age ≥18 years and < 65 years
* willingness to participate in this observational study
* minimum disease duration of 5 years
* brittle diabetes, as defined by the occurrence of frequent acute complications (ketoacidosis or severe hypoglycaemic episodes requiring third-part assistance or unawareness despite well-conducted intensive insulin therapy)
* presence of at least one diabetes-related complication (either neuropathy, retinopathy, subclinical nephropathy).

Exclusion Criteria (both groups)

* conditions other than T1D known to affect bone health (i.e., non-compensated hypothyroidism, hyperthyroidism, hyperparathyroidism, inflammatory bowel disease, malignancy, rheumatoid arthritis, hypogonadism, severe chronic obstructive pulmonary disease, hepatic insufficiency, alcohol intake ≥ 3 units/day ),
* use of drugs that can affect bone metabolism (e.g., bisphosphonates, anticonvulsants, hormone replacement therapy) other than glucocorticoids and immunosuppressants
* recipients of simultaneous pancreas kidney transplantation, pancreatic islet transplantation, multiple PTAs, other transplants
* BMI <18.5 or ≥ 30 kg/m2

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: All patients who underwent their first deceased donor PTA, or second deceased donor PTA if their first graft was explanted within a week, at the IRCCS San Raffaele Hospital between 2 January 2005 and 31 December 2017 will be screened for this study. Controls will be selected among outpatients with T1D attending the Endocrinology Unit at IRCCS San Raffaele Hospital and those listed for a first deceased donor PTA.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Fracture incidence | 02 January 2005 - 30 September 2018
  Difference in fracture incidence (any fracture) between the PTA and the control group

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Scientific Institute, Milan, Please Select, Italy